CLINICAL TRIAL: NCT07161804
Title: A Single-blind Randomized Placebo Controlled Pilot Study With Individualized Homeopathic Treatment in the Children With Autism Spectrum Disorder (ASD)
Brief Title: Pilot RCT Using Homeopathic Medicines in ASD
Acronym: Pilot-RCT-ASD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holistic Homoeopathic Clinic and Research Center (Other)
Responsible Party: Principal Investigator, Gyandas Wadhwani, Principal Investigator, Holistic Homoeopathic Clinic and Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201724112024
Record Dates: First submitted 2025-07-27; First posted 2025-09-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: ASD; RCT; HOMEOPATHY
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Homeopathy; Dosage Forms; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homoeopathic Group (Experimental): Individualized Homoeopathic Medicines
  Interventions: Drug: Homoeopathic medicines; Behavioral: Therapy
- Control Group (Placebo Comparator): Placebo
  Interventions: Behavioral: Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Homoeopathic medicines — Thuja officinalis Vaccininum Causticum Argentum nitricum Tuberculinum Stramonium Staphysagria Arum triphyllum Bacillinum Cina Carcinocin Cuprum Metallicum Ambera grisea Calcarea carbonica Crocus sativus Hepar sulphur Hyoscymus Kali Bromatum Lac Vaccininum Medorrhinum Natrum phosphoricum Thyroidinum
  Other Names: Medicines
  Arms: Homoeopathic Group
Behavioral: Therapy — Occupational Therapy / Speech Therapy
Drug: Placebo — Saccharum lactis
  Arms: Control Group

SUMMARY:
This study looked at whether homeopathic treatment could help children with Autism Spectrum Disorder (ASD) when used alongside regular therapies like speech and occupational therapy. Over seven years, children between the ages of 3 and 12 were divided into two groups (through computer generated list). One group received individualized homeopathic medicines, and the other received a look-alike placebo (with no active ingredients). Meanwhile, both the groups continued with their regular therapies.

Researchers used various tools and parent questionnaires to track the children's progress in areas like communication, behavior, social skills, daily functioning, toilet training and sensory skills.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are lifetime neurodevelopmental disorders with challenges across functional domains. Despite availability of various treatment modalities and diagnostic tools, it's pathophysiology still remains poorly understood even through 8 decades of it's discovery. This pilot study compares psychometrics and parental reported outcome monitoring, behavioral and developmental outcomes, co-occurring breadth of concerns for children with ASD along with co-morbidities, with and without homeopathic treatment.

Methodology: Initial screening was done using Autism Behavior Checklist (ABC). Utilizing a randomized-controlled design and parental informed consent, this study compared children aged 3 to 12 years, divided into an experimental group receiving individualized homeopathic treatment alongside occupational/speech therapies (HG), and a control group receiving only latter (CG) .

The treatment group received homoeopathic medicines daily with frequency being once per day along with daily occupational / speech therapy sessions for 1 hour each. The control group received homoeopathic medicine look alike placebo daily with frequency being once per day along with daily occupational / speech therapy sessions for 1 hour each. Follow ups were done every 3 months and the data were combined and stored for each year separately for seven-years. The data was initially collected and then analyzed through standardized behavioral assessments [Childhood Autism Rating Scale, CARS] , speech-language assessments [Social Responsiveness Scale, SRS], parental-questionnaires for reporting emotional regulation, anxiety-related behaviors, co-morbidities [Neuro Developmental Parent Report for Outcome Monitoring, ND-PROM] and observational methods in both the groups. The treatment effectiveness was assessed using Autism Treatment Evaluation Checklist (ATEC).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of Autism Spectrum Disorder (ABC score ≥ 67)
* Age range of 2 to 12 years

Exclusion Criteria:

* Children with other significant comorbid psychiatric conditions that could confound the results. [eg. a brain injury; fragile X syndrome or other syndromes resulting from known genetic defects or inherited metabolic diseases; other diagnosed conditions involving impairments in social and communication abilities, such as intellectual disability without ASD, global developmental delay, language disorders and social communication disorder]
* Children with irregular follow ups.
* Children with poor medical compliance.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | Baseline, Yearly (0 - 7 years)
  To measure various behavioral dimensions and adaptive functioning
Autism Treatment Evaluation Checklist (ATEC) | Baseline, Yearly (0 - 7 years)
  To assess the efficacy of the treatment among both the arms.

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | Baseline, Yearly (0 - 7 years)
  To measure social skills, communication abilities.
Neurodevelopmental Parent Report for Outcome Monitoring (ND PROM) | Baseline, Yearly (0 - 7 years)
  To gather subjective reports on their children's behavior, social interactions, and overall well-being from the parents.

CONTACTS AND LOCATIONS:
Overall Officials: GYANDAS G WADHWANI, MD (HOM.), Principal Investigator — Holistic Homoeopathic Clinic and Research Center
Locations (1):
- Holistic Homoeopathic Clinic and Research Center, New Delhi, SOUTH DELHI, India

IPD SHARING:
Plan to Share IPD: No
TO MAINTAIN CONFIDENTIALITY